CLINICAL TRIAL: NCT04972357
Title: Bariatric Procedures and Changes in Gut Hormone and Gastric Passage
Brief Title: Bariatric Procedures and Changes Gastric Passage
Acronym: BIP
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1172
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Gastric Emptying; Roux-en-Y Gastric Bypass; Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard RYGB
- Banded RYGB
- Extended pouch RYGB

SUMMARY:
Gastric emptying measured with scintigraphy in patients after standard Roux-en-Y Gastric Bypass (S-RYGB), Banded-RYGB (B-RYGB) or Extended pouch-RYGB (E-RYGB).

ELIGIBILITY:
Inclusion Criteria:

Female patients who underwent S-RYGB, B-RYGB or E-RYGB as a primary bariatric surgery.

Exclusion Criteria:

(1) had a disease known to affect appetite, gastric emptying or gastrointestinal motility (e.g., diabetes mellitus or hyper-/hypothyroidism); (2) were unable to stop medications that affect gastric emptying and/or motility three days prior to measurements (e.g., anti-cholinergic drugs, prokinetics, theophylline, calcium blocking agents, opioids); (3) started menopause; (4) were pregnant or lactating; (5) had a drug or alcohol addiction; (6) were unable to stop smoking for 24 hours.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Female patients who inderwent S-RYGB, B-RYGB or E-RYGB as a primary bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | cross-sectional study. Measured once over a period of 45-60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided